CLINICAL TRIAL: NCT01994486
Title: Open-Label Study to Evaluate the Safety and Tolerability of Telaprevir in Combination With Sofosbuvir in Treatment Naive Subjects Chronically Infected With Hepatitis C Virus Genotype 1
Brief Title: Open-Label Safety Study of Telaprevir and Sofosbuvir in Chronic Hepatitis C Genotype 1
Acronym: STEADFAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20132125
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis C, Chronic
Keywords: HCV Genotype 1; Hepatitis C Virus Genotype 1; HCV; TVR
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telaprevir and Sofosbuvir (Experimental): All subjects will receive Telaprevir twice a day, 1125mg capsule and Sofosbuvir 400 mg capsule once daily. Both will be given for 12 weeks.
  Interventions: Drug: Telaprevir and Sofosbuvir

INTERVENTIONS:
Drug: Telaprevir and Sofosbuvir — All subjects will have time to read and discuss IRB approved consent form prior to any study procedures. Following proper consenting, subjects will undergo physical exam including ECG and bloodwork prior to baseline visit. Subjects will return for research visits (vitals, collection of AEs, bloodwork, drug accountability) on Day 3, Weeks 1, 2, 3, 4, 6, 8, 10 and 12 of treatment and 4, 12, and 24 weeks after end of treatment. PK samples will be collected at week 2 and week 10.
  Other Names: TVR; SOF

SUMMARY:
This is an open-label, multi center study of treatment-naive non-cirrhotic subjects with genotype 1 chronic Hepatitis C Virus. All subjects will receive telaprevir (TVR) in combination with sofosbuvir (SOF) for 12 weeks.

DETAILED DESCRIPTION:
Starting on Day 1 and for up to 12 weeks, you will receive Telaprevir (TVR) and Sofosbuvir (SOF).

You will take one (1) 400 mg tablet of SOF and 3 tablets (1125 mg each) of TVR. You should take these together by mouth every morning. You will take another 3 tablets (1125 mg each) of TVR by mouth 12 hours after you take your morning dose.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* BMI (Body Mass Index) ≥ 18 kg/m2
* HCV RNA quantifiable at screening and >1,000 IU/ml
* HCV treatment Naïve
* HCV genotype 1
* 7. Confirmation of chronic HCV infection documented by either: A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or A liver biopsy performed prior to the Baseline/Day 1 visit with evidence of chronic HCV infection

Exclusion Criteria:

* Current or prior history of any of the following:

Clinically-significant illness Cirrhosis 2. Screening ECG with clinically significant abnormalities

1. ALT > 10 x the upper limit of normal (ULN)
2. AST > 10 x ULN
3. Direct bilirubin > 1.5 x ULN
4. Platelets < 150,000/μL
5. HbA1c > 7.5%
6. Creatinine clearance (CLcr) < 60 mL /min, as calculated by the Cockcroft-Gault equation
7. Hemoglobin < 11 g/dL for female subjects; < 12 g/dL for male subjects.
8. Albumin < 3.1 g/dL
9. INR > 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR 4. Prior exposure to any approved or experimental HCV-specific direct-acting

   5. Pregnant or nursing female or male with pregnant female partner.

   6. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, cholangitis).

   7. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DAVID R NELSON, MD, Study Director — University of Florida
Locations (1):
- UF Hepatology Research at CTRB, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Telaprevir and Sofosbuvir: All subjects will receive Telaprevir 1125 mg capsule twice a day with Sofosbuvir 400 mg capsule once daily for 12 weeks.
  In addition, sparse PK samples will be collected at week 2 and week 10.
Period: Overall Study
Arm/Group | Telaprevir and Sofosbuvir
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: HCV GENOTYPE 1 -NON-CIRRHOTIC ADULTS
Groups:
- Telaprevir and Sofosbuvir: All subjects will receive Telaprevir twice a day, 1125mg capsule and Sofosbuvir 400 mg capsule once daily. Both will be given for 12 weeks.
  Telaprevir and Sofosbuvir: All subjects will have an ECG performed. Then they will receive Telaprevir twice a day, 1125mg capsule and Sofosbuvir 400 mg capsule once daily. Both will be given for 12 weeks. In addition, PK samples will be collected at week 2 and week 10.
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 51 [20 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events Leading to Discontinuation of Both Telaprevir and Sofosbuvir Among Subjects Treated With Telaprevir and Sofosbuvir
Description: Study drug adherence and adverse events were collected on all enrolled subjects and graded using the DAIDS scale. Any adverse events leading to discontinuation of both Telaprevir and Sofosbuvir were collected and are hereby reported.
Time Frame: 12 weeks-January 3, 2014- April 10, 2014
Population: Non-cirrhotic Hepatitis C Genotype 1 infected subjects, naive to previous Hepatitis C treatment
Measure: Number; unit: participants
Groups:
- Telaprevir and Sofosbuvir: All subjects will receive Telaprevir twice a day, 1125mg capsule and Sofosbuvir 400 mg capsule once daily for 12 weeks.
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Characterize Steady State of Sofosbuvir Active SOF Metabolite, GS-331007
Description: Sparse Pharmokinetic blood samples were collected at Week 2 and Week 10 (prior to daily dose) in patients treated with Telaprevir and Sofosbuvir.
Time Frame: 1/17/2014-3/26/2014
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
ng/mL
  Pre-Dose Trough Level Metabolite GS-331007 Wk 2 | 593 (181)
  Pre-Dose Trough Level GS-331007 Wk 10 | 619 (216)

3. Other Pre Specified Outcome: Number of Subjects With Sustained Virologic Response at 4 Weeks After Completion of Last Dose
Description: Subjects who complete assigned treatment and have undetectable HCV RNA at 12 weeks after the last planned dose of study treatment
Time Frame: 4/22/2014-5/6/2014
Measure: Number; unit: participants
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
participants | 19

4. Secondary Outcome: Proportion of Subjects Who Achieve Undetectable Hepatitis C Virus RNA at 12 Weeks After Completing Study Drug Regimen
Description: Plasma HCV RNA levels were assessed using the COBAS TaqMan HCV RNA assay test (v2.0; Roche Diagnostics, Indianapolis, IN, USA; LLOQ=25 IU/mL;limit of detection =15 IU/mL)
Time Frame: 6/16/2014-7/2/2014
Measure: Number; unit: participants
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
participants | 19

5. Primary Outcome: Safety of Telaprevir and Sofosbuvir When Dosed in Combination for 12 Weeks
Description: The number of subjects who experienced Grade 3 anemia. Complete blood count was collected at baseline, week 2, week 4, week 8, week 12, week 18, and week 24. Incidence of moderate anemia (Grade 3) observed in the study treatment period.
Time Frame: 1/3/2014-4/10/2014
Measure: Number; unit: participants
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
participants | 1

6. Secondary Outcome: Proportion of Subjects With Viral Relapse
Description: Defined as Subjects who have undetectable HCV RNA at end of treatment, and confirmed detectable HCV RNA between end of treatment and SVR12 planned assessment time point.
Time Frame: 1/3/2014-9/8/2014
Measure: Number; unit: participants
Arm/Group | Telaprevir and Sofosbuvir
Number analyzed (Participants) | 20
participants | 1

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: AEs collected from all subjects beginning at baseline through 28 days after last dose of study medication were assigned to treatment phase for evaluation.
Arm/Group | Telaprevir and Sofosbuvir
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telaprevir and Sofosbuvir (N=20)
Bradycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telaprevir and Sofosbuvir (N=20)
Abdominal bloating (Gastrointestinal disorders) | 1 (1)
Abdominal cramps (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Anorectal_symptoms (Gastrointestinal disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Flushing (Vascular disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Head cold (Infections and infestations) | 2 (3)
Head pressure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperactivity (Psychiatric disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Increased frequency of bowel movements (Gastrointestinal disorders) | 1 (1)
Induration (General disorders) | 2 (3)
Irritability (General disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral edema (General disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Regurgitation (Gastrointestinal disorders) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tingling (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No